CLINICAL TRIAL: NCT04440488
Title: A Prospective, Randomized, Double-Blind, Parallel Group Study to Evaluate the Safety and Efficacy of ARALAST NP 60 mg/kg and 120 mg/kg for Alpha-1 Proteinase Inhibitor (A1PI) Augmentation Therapy in Subjects With A1PI Deficiency and Chronic Obstructive Pulmonary Disease-Emphysema (COPD-E)
Brief Title: ARALAST NP Alpha-1 Lung Density Chronic Obstructive Pulmonary Disease-Emphysema (COPD-E) Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Reevaluation of development strategy
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-883-3001
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARALAST NP 120 mg/kg (Experimental): Participants will receive 120 mg/kg BW of ARALAST NP intravenous (IV) infusion once in a week for a total of 104 weeks which will be compared with an external placebo arm.
  Interventions: Biological: ARALAST NP
- ARALAST NP 60 mg/kg (Experimental): Participants will receive 60 mg/kg BW of ARALAST NP IV infusion once in a week for a total of 104 weeks which will be compared with an external placebo arm.
  Interventions: Biological: ARALAST NP

INTERVENTIONS:
Biological: ARALAST NP — Partcipants will be randomized to receive ARALAST NP 60 or 120 mg/kg BW/week IV infusion for a total of 104 weeks.
  Other Names: Alpha1-PI; TAK-883; A1PI; Alpha1-Proteinase Inhibitor (Human)

SUMMARY:
The purpose of this study is to evaluate the efficacy of ARALAST NP A1PI augmentation therapy 120 milligrams per kilogram (mg/kg) body weight (BW)/week compared with an external placebo comparator on the loss of emphysematous lung tissue measured by lung density change in participants with A1PI deficiency and COPD-E.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years of age at the time of screening
* Diagnosis of A1PI deficiency with endogenous plasma A1PI level less than (<) 11 micromoles(μM) (< 0598 milligram per milliliter [mg/mL]) following 4-week minimum washout from previous last dose of A1PI augmentation therapy The screening plasma A1PI level may be repeated if a participant is determined to have an exclusionary value that maybe due to an inadequate washout of augmentation therapy Participants eligible for enrollment include newly diagnosed, previously untreated, currently treated and currently not on treatment but received treatment in the past
* Participants should have a documented A1PI genotype and if not, A1PI genotyping will be offered at the time of screening The purpose for genotyping is for sub-group analysis of study results only
* Clinically evident COPD-E (according to GOLD criteria (2020) for diagnosis, Stage I-III) (Global Initiative for Chronic Obstructive Lung Disease [COPD]) at the time of screening defined as follows: Forced expiratory volume in 1 second (FEV1) is greater than or equal to (>or=) 35% and less than or equal to (<or=) 70% predicted
* If treated with any respiratory medications including inhaled bronchodilators, inhaled corticosteroids, or systemic corticosteroids (example [eg] prednisone <or= 10 milligram per day [mg/day] or its equivalent), the doses of medications should have remained stable for at least 28 days prior to screening
* No clinically significant abnormalities (other than emphysema, bronchitis or bronchiectasis) detected via chest CT at the time of screening
* Males and non-pregnant, non-lactating females whose screening pregnancy test is negative and willing and able to employ adequate contraceptive methods deemed reliable by the investigator for the duration of the study
* Willing and able to refrain from smoking (including e-cigarettes and vaping of any other substance) for the duration of study
* Willing and able to comply with the requirements of the protocol and able to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) an informed consent to participate in the study

Exclusion Criteria:

* Known ongoing or history of clinically significant disease other than respiratory or liver disease secondary to AATD
* If experiencing corona virus diease (COVID)-19, lower respiratory tract infection (LRTI) and/or acute COPD exacerbation at the time of screening. Participant may be re-screened after clinical resolution of COVID-19, LRTI and/or acute COPD exacerbation and having also remained stable for at least 6 weeks after resolution
* Known ongoing or history of clinically significant cor pulmonale and/or congestive heart failure with New York Heart Association (NYHA) Class III/IV symptoms
* Has received an organ transplant, has undergone major lung surgery (eg, lung volume reduction surgery or lobectomy surgery), or is currently on a transplant waiting list
* Known history of ongoing malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, or stable prostate cancer not requiring treatment)
* Current active smoker (including e-cigarettes or vaping, nicotine or any other substance). A participant with a previous history of smoking has to have ceased active smoking at least 6 months prior to screening. Participants with a positive nicotine/cotinine test due to nicotine replacement therapy (eg, patches, chewing gum) or snuff are eligible
* Receiving long-term therapy (> 28 days) of parenteral corticosteroids or oral corticosteroids at doses greater than 10 mg/day of prednisone or its equivalent
* Receiving chronic 24 hours/day oxygen supplementation (other than for an acute COPD exacerbation, or supplemental oxygen with continuous positive airway pressure [CPAP], or bi-level positive airway pressure [BiPAP] for acute respiratory failure)
* Known selective immunoglobulin A (IgA) deficiency (IgA level < 7 milligrams per deciliter [mg/dL] at screening) with anti-IgA antibodies and a history of hypersensitivity reaction
* Known history of hypersensitivity following infusions of human immunoglobulins, human albumin, blood or blood components
* Presence of clinically significant laboratory abnormalities at the screening that in the opinion of the investigator would impact the participant's safety, if enrolled in the study
* Presence of any of the following that in the opinion of the investigator, would affect participant's safety or compliance or confound the results of the study, including known clinically significant medical, psychiatric, or cognitive illness, is a recreational drug/alcohol user, or has any other uncontrolled medical condition (eg, unstable angina, transient ischemic attack, uncontrolled hypertension)
* Known exposure to another IP within 28 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
* Participant is a family member or employee of the investigator
* If female, participant is pregnant or nursing at the time of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-08 (Estimated); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Annual Rate of the Physiologically Adjusted Lung Density Change | Baseline, up to Week 104
  Annual rate of the physiologically adjusted lung density change will be measured as the 15th percentile of the lung density measurements (PD15) as assessed by Computed Tomography (CT) densitometry at total lung capacity (TLC). CT lung density at the 15th percentile (PD15) is the threshold below which 15 percentage (%) of the voxels have lower densities and is used as the parameter for estimating the rate of lung density decline. Annual rate of the physiologically adjusted lung density change will be tested in a fixed comparision sequence 1. ARALAST NP 120 mg/kg BW/week group versus (vs) external placebo group, 2. ARALAST NP120 mg/kg BW/week vs 60 mg/kg BW/week, 3. ARALAST NP 60 mg/kg BW/week group vs external placebo group.

SECONDARY OUTCOMES:
Number of Moderate or Severe Exacerbations of Chronic Obstructive Pulmonary Disease (COPD) | Baseline, up to Week 104
  COPD exacerbations are defined as an acute worsening of respiratory symptoms that results in additional therapy and will be assessed according to the classification in GOLD criteria (2020) as follows: Moderate (treated with short acting bronchodilators [SABDs] plus antibiotics and/or oral corticosteroids) and Severe (required hospitalizations or a visit to the emergency room).
Annual Rate of Change in Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) | Baseline, up to Week 104
  Annual rate of change in post-bronchodilator FEV1 will be assessed.
Number of Participants with Treatment-Emergent Adverse Events (TEAE's) | From Start of the study drug administration up to End of the study (up to Week 105)
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this IP or medicinal product. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. TEAE's will include related, serious adverse events (SAEs), suspected adverse reactions plus adverse reactions of interest, temporally-associated adverse events (AEs) with onset during infusion or within 24 hours following the end of IP infusion, and AEs resulting in changes to infusion dose.
Number of Participants Who Develop Anti-A1PI Antibodies Following Treatment With ARALAST NP | From Start of the study drug administration up to End of the study (up to Week 105)
  Number of participants who develop anti- A1PI antibodies following treatment with ARALAST NP will be assessed.
Plasma Trough Level of Antigenic and Functional A1PI for ARALAST NP at each dose Level | Pre-dose, Weeks 4, 13, 28, 52, 78, 91, 104, 105
  Plasma trough level of antigenic and functional A1PI for ARALAST NP at each dose level (ARALAST NP 60 mg/kg BW/week, ARALAST NP 120 mg/kg BW/week) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire

IPD SHARING:
Plan to Share IPD: Yes
Shire provides access to the de-identified individual participant data for eligible studies to aid qualified researchers in addressing legitimate scientific objectives. These IPDs will be provided following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.shiretrials.com website. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://www.shiretrials.com/en/our-commitment-to-transparency/data-sharing-with-researchers